CLINICAL TRIAL: NCT05454241
Title: Efficacy, Safety and PK of CD7 CAR-T in Patients With Relapsed or Refractory CD7+ Hematological Malignancies
Brief Title: CD7 CAR-T for Patients With r/r CD7+ Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022020
Record Dates: First submitted 2022-07-04; First posted 2022-07-12 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2023-06

CONDITIONS: Hematological Malignancies
Keywords: T-ALL/LBL; AML
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD7 UCAR-T cells (Experimental)
  Interventions: Drug: Anti-CD7 CAR-T

INTERVENTIONS:
Drug: Anti-CD7 CAR-T — Universal CAR-T cells targeting CD7

SUMMARY:
This is a open-label, phase 2 study to evaluate the efficacy, safety and PK of CD7 chimeric antigen receptors treatment for patients with refractory/relapsed CD7 positive hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed CD7 positive relapsed/refractory hematological malignancies.
2. Echocardiography shows left ventricular ejection fraction (LVEF) ≥ 50%;
3. There is no active pulmonary infection, and the oxygen saturation during air inhalation is more than 92%;
4. The estimated survival time is more than 3 months;
5. Eastern cooperative oncology group (ECOG) performance status of 0 to 2
6. The patients or their legal guardians voluntarily participated in the trial and signed the informed consent.

Exclusion Criteria:

1. Patients with history of epilepsy or other central nervous system diseases;
2. Patients with prolonged QT or severe heart disease;
3. Pregnant or lactating women
4. Patients with uncontrolled active infection.
5. Positive for any of the following etiological tests: HIV, HBV, HCV
6. Any other conditions that researcher think it is inappropriate for the subject to anticipate the trial

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | 1 Year
  Number of patients who achieved response after treatment of CD7 CAR-T cell.

SECONDARY OUTCOMES:
Duration of overall response (DOR) | 1 Year
  Duration of overall response will be assessed from the CAR-T cell infusion to progression, death or last follow-up.
Overall survival(OS) | 1 Year
  OS will be assessed from the CAR-T cell infusion to death or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Dr., Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No
When the research is completed, it will be shared in the form of a paper publication